CLINICAL TRIAL: NCT03262415
Title: PRECISION Study: Evaluating the Accuracy of the LabPatch Continuous Glucose Monitor
Status: Completed | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Cambridge Medical Technologies, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CHS #: 2016-31
Record Dates: First submitted 2017-08-17; First posted 2017-08-25 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Type1 Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: LabPatch Continuous Glucose Monitoring (CGM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 20 to 22 blood sample( A total of about 110 mL of blood will be drawn during the visit).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: 30 adult subjects with type 1 or type 2 diabetes treated with insulin. The accuracy of the LabPatch Continuous Glucose Monitoring (CGM) will be evaluated during the study visit, comparing to YSI 2300 STAT Plus, OneTouch Verio and FreeStyle Lite.
  Interventions: Device: LabPatch Continuous Glucose Monitoring (CGM)

INTERVENTIONS:
Device: LabPatch Continuous Glucose Monitoring (CGM) — 1. The patch device that will be applied to subjects' arms in this study is about 3 inches in length and one inch in width, with adhesive tape on the sides.
  2. The LabPatch circuit chip lies on the underside of the bandage. The circuit is in the form of a small chip (approximately 15.7 mm [0.618"] x 15.7 mm [0.618"]) placed in contact with the skin. The chip has a telescopic micropipette which draws interstitial fluid to be analyzed for glucose levels. The chip is also able to measure skin temperature to ensure appropriate skin contact.
  3. A wire that connects the chip to a laptop that continuously captures glucose data.

SUMMARY:
The purpose of this study is to evaluate the accuracy and efficacy of the Cambridge Medical Technologies, LLC LabPatch Continuous Glucose Monitoring (CGM) System compared to a laboratory glucose analyzer (YSI 2300 STAT Plus) and 2 commercial glucometers, OneTouch Verio and Freestyle Lite.

The LabPatch system includes:

1. The LabPatch circuit chip which lies in the center of a circular push-button. The circuit is in the form of a small chip (approximately 15.7 mm [0.618"] x 15.7 mm [0.618"]) placed in contact with the skin. The chip has a telescopic micropipette which draws interstitial fluid to be analyzed for glucose levels. The chip is also able to measure skin temperature to ensure appropriate skin contact.
2. A Lab Patch holding device (blue box).
3. A wire that connects the chip to a laptop that continuously captures glucose data.

DETAILED DESCRIPTION:
Study design:

This is a cross-sectional, pilot, precision, single center, single-arm study, enrolling 30 adult subjects with type 1 or type 2 diabetes treated with insulin.

The study will include both a screening visit and a single study visit.The accuracy of the LabPatch CGM will be evaluated during the study visit, comparing to YSI 2300 STAT Plus, OneTouch Verio and FreeStyle Lite.

Screening Visit:

Following the informed consent process, screening evaluation will determine subject eligibility for enrollment, including:

* Demographics- including age, sex at birth, race/ethnicity, dominant hand, and BMI.
* Diabetes History - including type of diabetes, date of diagnosis or length of diabetes, history of DKA and severe hypoglycemia, current treatment [type of insulin and type of insulin delivery (injections or insulin pump)], insulin doses, and when applicable: basal rates, correction factors, glucose targets, insulin duration, insulin to carbohydrate ratios, sliding scales.
* Current and Past Medical History - including current medications.
* Physical examination and vital signs- including height, weight, blood pressure, pulse, assessment of venous access for repeated blood draws.

Study Visit (visit window: screening visit + 0 to 30 Days):

Subject Admission

The subject will arrive at the clinical research center at Joslin Diabetes Center during the day, no later than 10:00 AM and the following will be performed:

* The study team will confirm the absence of fever, nausea or vomiting that might occur within 24 hours before the visit.

During this visit the following procedures will be conducted:

* Measurement of BP and anthropometric parameters will be taken and include, weight, height and BMI.
* An intravenous line will be inserted through which all blood samples will be collected.
* The study team will prepare the sensor and its connectors appropriately.
* A fasting blood sample will be collected for measurement plasma glucose, A1C and complete blood count.
* A breakfast meal will be given followed 3-4 hours later by a lunch.
* Insulin will be injected before breakfast and lunch based on the blood glucose value before the meal using the same insulin regimen by the subject in the outpatient setting.
* At 15 minute intervals, subject will sit down at a mobile "overbed" table that has the LabPatch CGM. Then, they will press with their major finger on a circular push-button for about 15 seconds for each measurement of glucose. When pressed, the LED ring light illuminates in blue, indicating that the glucose measurement has commenced. The finger will remain in place until a beep is heard, then lifted.
* Twenty to 22 blood samples will be drawn during the study visit. The samples will be drawn at the following intervals: baseline, every 15 minutes for 2 hours after breakfast, every 30 minutes till the lunch time, and every 15 minutes for 2 hours after lunch. A total of about 110 mL of blood will be drawn during the visit.
* If all admission criteria are not met, the subject will be rescheduled. If all of the admission readiness conditions are met, the subject will be admitted to the Clinical Research Center (CRC).

Before discharge:

* Finger-stick glucose will be assessed.
* If plasma glucose is <70 mg/dL, 15 gm of carbohydrates will be given to raise the glucose to ≥100 mg/dL and blood glucose will be checked after 15 min and another carbohydrates dose is given if blood glucose is still <70 mg/dL. Subject will be only allowed to go home when the blood glucose is >100 mg/dL and stable.

Subject Instructions prior to the visit

* Prior to admission, subjects should check their blood glucose, if it is <70 mg/dL or subject feels hypoglycemic symptoms, then they should eat a snack prior to coming to the visit

Estimated Visit Duration

* The total duration of the inpatient visit is approximately 6 hours with screening visit being approximately 2 hour. The study time may be extended for glucose stabilization prior to discharge.

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board/Independent Ethics Committee, and provided Health Insurance Portability and Accountability Act authorization (HIPAA) or other privacy authorization prior to any participation in study.
* Subject is between 18 and 75 years of age.
* Subject is diagnosed with type 1 diabetes for ≥3 months and is being treated with insulin injections in the form of multiple daily injections or through insulin infusion pump.
* Subject is diagnosed with type 2 diabetes for ≥3 months and is being treated with insulin in the form of multiple daily injections or through insulin infusion pump.
* Subject is a male or a non-pregnant and non-lactating female, at least 6 weeks postpartum prior to screening visit. A urine pregnancy test is required for all female subjects unless she is not of childbearing potential, defined as postmenopausal for at least one year prior to screening visit or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

* Subject is pregnant or lactating.
* Subject is not treated with insulin.
* Subject has/had acute or chronic, contagious, infectious disease
* Subjects with history of blood-born chronic viral infection (e.g. Hepatitis C and HIV)
* Subject has/had clotting or bleeding disorders or other hematological disease.
* Subject has an active malignancy (excluding the following dermal malignancies: basal cell carcinoma, squamous cell carcinoma, carcinoma in-situ of the cervix).
* Subject had a recent cardiovascular event (e.g., myocardial infarction, stroke) ≤ six months prior to screening visit; or stated history of congestive heart failure.
* Subject has known allergy to adhesive material present in commercial bandages

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with type 1 or type 2 diabetes treated with insulin.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Mean absolute relative difference (MARD) | Baseline, every 15 minutes after breakfast for 2 hours, every 30 minutes until lunch time, and every 30 minutes after lunch for 2 hours
  Blood glucose values (mg/dL) from the LabPatch system and reference YSI, One Touch Verio, and FreeStyle Lite will be used to report the mean absolute relative difference (MARD) in Percentage (%).

CONTACTS AND LOCATIONS:
Overall Officials: Osama Hamdy, M.D.,Ph.D, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No